CLINICAL TRIAL: NCT00332488
Title: A Phase 3, 24-Week, Multi-Center, Open-Label, Randomized, Controlled Trial Comparing the Efficacy and Safety of Prandial Inhalation of Technosphere/Insulin in Combination With Metformin or Technosphere/Insulin Alone Versus 2 Oral Anti-Diabetic Agents (Metformin and a Secretagogue) in Subjects With Type 2 Diabetes Mellitus Sub-optimally Controlled on Combination Metformin and a Secretagogue.
Brief Title: Efficacy and Safety of Prandial Inhalation of Technosphere/Insulin in Combination With Metformin or Technosphere/Insulin Alone Versus 2 Oral Anti-Diabetic Agents in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-103
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Secretagogues

ARMS (3):
- 1 (Experimental): Technosphere Insulin
  Interventions: Drug: Technosphere Insulin
- 2 (Active Comparator): Metformin & Secretagogues
  Interventions: Drug: Metformin & Secretagogues
- 3 (Experimental): Technosphere & Metformin
  Interventions: Drug: Technosphere Insulin & Metformin

INTERVENTIONS:
Drug: Technosphere Insulin — Inhalation, 15U/30U, prandial
  Arms: 1
Drug: Metformin & Secretagogues — Metformin tablets,Secretagogues supplied as any of the currently marketed brands and formulations.
  Arms: 2
Drug: Technosphere Insulin & Metformin — Technosphere Insulin Inhalation Powder 15U/30U, Metformin tablets
  Arms: 3

SUMMARY:
to demonstrate the efficacy of inhaled Technosphere/Insulin in combination with metformin versus combination metformin and a secretagogue

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers with clinical diagnosis of Type 2 diabetes mellitus for >or= to 6 months
* Stable regimen of metformin for > or = to 1000mg/day or maximum tolerated dose) and a secretagogue < or = 1/2 the maximum manufacturer-recommended daily dose without any dose adjustments within the preceding 6 wks.
* Fixed dose combination products of metformin and sulfonylurea are acceptable as long as each individual dose meets inclusion criteria
* HbA1c >or= to 7.5% and < or= to 11.0%
* BMI < or = to 40kg/m2.
* FEV1> or = to 70%, Total Lung capacity and > or =80% DLco > or= to 70%

Exclusion Criteria:

* Treatment with any type of anti-diabetic therapy, other than metformin & secretagogues within the preceding 12 weeks
* Serum creatinine > 1.4mg/dL in female subjects and >1.5mg/dL in male subjects
* History of chronic obstructive pulmonary disease, clinically proven asthma and/or any other clinically important pulmonary function testing and/or radiologic findings
* Evidence of serious complications of diabetes (e.g. autonomic neuropathy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2004-12; Primary Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: For MannKind sponsored trials, the Overall Study Official is the Chief Scientific Officer, Study Director — Mannkind Corporation
Locations (120):
- United States (43):
  - Radiant Research-Birmingham, Birmingham, Alabama
  - Parkway Medical Center, Birmingham, Alabama
  - Redpoint Research, Phoenix, Arizona
  - Arizona Center for Clinical Research, Phoenix, Arizona
  - International Clinical Research Network, Chula Vista, California
  - National Jewish Medical & Research Center, Denver, Colorado
  - Creekside Endocrine Associates, Denver, Colorado
  - Jennifer Hone MD, Denver, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Center for Diabetes & Endocrine Care, Hollywood, Florida
  - International Research Associates LLC, Miami, Florida
  - Cedar-Crosse Research Center, Chicago, Illinois
  - John H Stoger Jr Hospital of Cook County, Chicago, Illinois
  - Clintell Inc, Skokie, Illinois
  - James A Dicke MDPA, Towson, Maryland
  - East Coast Clinical Research Inc, Haverhill, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Michigan Institute of Medicine, Livonia, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Clayton Medical Research, St Louis, Missouri
  - Raidant Research-St Louis, St Louis, Missouri
  - Creighton Diabetes Center, Omaha, Nebraska
  - Lovelace Scientific Resources (Albuquerque), Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Metrolina Internal Medicine, Charlotte, North Carolina
  - Charlotte Clinical Research Inc, Charlotte, North Carolina
  - Sensenbrenner Primary Care, Charlotte, North Carolina
  - Duke Medical Center, Durham, North Carolina
  - Dayton Clinical Research, Dayton, Ohio
  - Providence Health Partners - Center of Clinical Research, Dayton, Ohio
  - Radiant Research, Portland, Oregon
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Collierville Medical Specialists, Collierville, Tennessee
  - Memphis Internal Medicine (Kathawala), Memphis, Tennessee
  - GoodLife Medical Center PLLC, Memphis, Tennessee
  - Baylor Endocrine Center, Dallas, Texas
  - Quality Assurance Research Center Inc, San Antonio, Texas
  - Clinical Trials of Texas Inc, San Antonio, Texas
  - Covenant Clinic Research, San Antonio, Texas
  - Diabetes & Glandular Disease Research Assoc PA, San Antonio, Texas
  - SAM Clinical Research Center, San Antonio, Texas
  - Cedar Research, Tacoma, Washington
- Argentina (5):
  - Hospital Interzonal de Agudos Pedro Fiorito, Avellaneda, Buenos Aires
  - Centro Endocrinologic Tiempo, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Cons Asoc de Endocrinologia, Buenos Aires
  - CIMeL, Buenos Aires
- Brazil (8):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Ccbr Brasil Centro de Analises e Pesquisas Clinicas Ltda, Rio de Janeiro
  - Hospital Guilherme Alvaro, Santos
  - CPClin-Centro de Pesquisas Clinicas, São Paulo
  - UNIFRSP, São Paulo
  - Hospital do Rim e Hipertensao, São Paulo
  - Instituto de Pesquisa Clinica e Medicina Avancada, São Paulo
- Canada (6):
  - Quest Clinical Trials, Markham, Ontario
  - Lifestyle Metabolism Center, Oakville, Ontario
  - Lifestyle Metabolism Center, Thornhill, Ontario
  - Lifestyle Metabolism Center, Toronto, Ontario
  - Trial Management Group Inc (Henein, Toronto, Ontario
  - Unimedico Management, Richmond Hill
- Chile (4):
  - Hospital Padre Alberto Hurtado, Santiago, Santiago Metropolitan
  - Hospital Clinico Pontificia Universidad Catolica de Chile, Santiago
  - Hospital del Salvador, Santiago
  - Instituto de Informacion de Tramiento y Educacion en Salud, Santiago
- Czechia (8):
  - Diabetologicka a interni ambulance, Ostrava-Kunčice, CZE
  - Institute for Clinical and Exp Medicine, Prague, CZE
  - University Hospital Na Bulovce, Prague, CZE
  - Interní a diabetologická Outpatient, Ostrava, Ostrava
  - Diabetologicka ambulance (Chmura), Ostrava
  - II interni klinika FN Kralovske Vinohrady, Prague
  - Endokrinologicky ustav, Prague
  - 3rd Medical Department General Faculty Hospital, Prague
- Mexico (6):
  - Instituto Mexicano de Investigacion, Mexico City, Durango
  - Hospital Universitario Dr Jose E Gonzalez, Monterrey, Nuevo León
  - Hospital Santa Engracia-CIMA, Garza García
  - Centro de Estudios en Diabetes, Mexico City
  - Hospital General de Mexico Servicio EndocrinologiaJefe Del Servicio, Mexico City
  - OCA-MIRC, Monterrey
- Poland (8):
  - Klinika Endocrinologii Diabetologii I, Bialystock, POL
  - NZOZ Specjalistyczny Osrodek Internistyczno - Diabetologiczny, Bialystok, POL
  - Katedra I Klinika Chorob Metabolicznych Collegium Medicum Uniwersytety Jagiellonskiego, Krakow, POL
  - Instytut Centrum Zdrowia (009) Matki Polki, Lodz, POL
  - Spzital Kolejowy imm Wlodzimierza Roeflera, Pruszków, POL
  - Oddzial Kliniczny Diabetologii (009) Kliniczny nr 1 im Norberta Barlickiego Uniwersytety Meycznego, Lodz
  - Centrum Leczenia Chorob cywilizacyjnych, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej VIVAMED, Warsaw
- Russia (13):
  - NHI Kemerovo Regional Clinical Hospital, Kemerovo, RUS
  - NI Principal Military Clinical Hospital n a academician N.N. Burdenko of the Ministry of Defense, Moscow, RUS
  - NEI HPE Moscow State University of Medicine and Dentistry of FAHSD City Clinical Hospital #70, Moscow, RUS
  - NI Endrocrinological Research Centre of RAMS In patient replacing technologies department, Moscow, RUS
  - NI Moscow Regional Scientific Research Clinical Institute na MF Vladimirsky, Moscow, RUS
  - St Petersburg NHI City Polytclinic #77 City Diabetological Center #4, Saint Petersburg, RUS
  - Central Medical Sanitary Unit #122, Saint Petersburg, RUS
  - St Petersburg NHI Municipal Multi-Speciality Hospital # 2, Saint Petersburg, RUS
  - TUV Medico-Military Academy, Saint Petersburg, RUS
  - NEI HPE Smolensk State Medical Academy of FAHSD RNHI Smolensk Regional Clinical Hospital, Smolensk, RUS
  - MHI Clinical Hospital for Emergency Care na NV Soloviev, Yaroslavl, RUS
  - NHI Yaroslavl Regional Clinical Hospital, Yaroslavl, RUS
  - NI Central Clinical Hospital of RAS, Moscow
- Spain (5):
  - Complejo Hospitalario Nuestra Senora de Valme, Seville, Andalusia
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Universitario de la Princessa, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Corporacion Sanitaria Parc Tauli Unidad de Endocrinologia, Sabadell
- Ukraine (14):
  - Bukovinian State Medical University Dept of Clinical Immun, Chernivtsy, UKR
  - Dniepropetrovsh State Medical Academy, Dniepropetrovsk, UKR
  - Donetsk State Medical University, Donetsk, UKR
  - Donetsk State Medical University (Chair of Immun Allergogoly & Endocrin), Donetsk, UKR
  - Railway Clinical Hospital on Donetsk Station, Donetsk, UKR
  - Chair Family Med of National Med University, Kiev, UKR
  - Institute of Endocrinology and Metabolism, Kiev, UKR
  - Ukr Scientifically Practical Centre of Endocrine Surgery, Kiev, UKR
  - Odessa State Medical University Dept of Gen Practice and Med Rehab, Odesa, UKR
  - Odessa Reg. Clinical Hosp Outpatient Department, Odesa, UKR
  - Odessa State Med Dept of Family Med and Gen Practice, Odesa, UKR
  - Vinnitsa State Medical University, Vinnitsa, UKR
  - Outpatient Clinic of Family Physician "Rusanovka", Kiev
  - Public Institution City Policlinic #20 Odessa, Odesa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 May 2006 (first subject enrolled) to 03 Mar 2008 (last subject completed. Multi-national trial conducted in Argentina, Brazil, Canada, Chile, Czech Republic, Mexico, Poland, Russian Federation, Spain, Ukraine, and USA.
Pre-assignment Details: 2 week screening period prior to randomization. 1512 patients screened with 528 patients randomized. 977 patients failed screening criteria, 9 subjects passed screening but were not randomized, 2 subjects failed screening but were randomized.
Groups:
- TI Inhalation Powder Alone: Technosphere® Insulin Inhalation Powder administered prior to each meal without any other anti-diabetic treatment; dose individualized for each subject
- Metformin & Secretagogues: Metformin (>= 1,000 mg/day or maximum tolerate dose) & Secretagogue (Sulfonylurea or meglitinide at >= half maximum manufacturer recommended dose or maximum tolerated dose)
- TI Inhalation Powder + Metformin: Technosphere® Insulin Inhalation Powder administered prior to each meal (dose individualized for each subject) & Metformin (>= 1,000 mg/day or maximum tolerate dose)
Period: Initial Treatment Phase (Weeks 0 - 12)
Arm/Group | TI Inhalation Powder Alone | Metformin & Secretagogues | TI Inhalation Powder + Metformin
Started | 183 | 170 | 175
Completed | 133 | 152 | 119
Not Completed | 50 | 18 | 56
Not completed — Adverse Event | 8 | 2 | 6
Not completed — Physician Decision | 13 | 2 | 10
Not completed — Withdrawal by Subject | 21 | 10 | 20
Not completed — Various | 4 | 0 | 20
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Protocol Violation | 3 | 1 | 0
Period: Transfer Treatment Phase (Weeks 12 - 24)
Arm/Group | TI Inhalation Powder Alone | Metformin & Secretagogues | TI Inhalation Powder + Metformin
Started | 29 (Subjects on TI who achieved an HbA1c < 7.5% or had an HbA1c decrease from baseline >= 1.0%) | 72 (Subjects on treatment who achieved an HbA1c < 7.5% or had an HbA1c decrease from baseline >= 1.0%) | 254 (Subjects in this arm who met HbA1c criteria + subjects from other arms who did not)
Completed | 27 | 70 | 233
Not Completed | 2 | 2 | 21
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 8
Not completed — Various | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TI Inhalation Powder Alone | Metformin & Secretagogues | TI Inhalation Powder + Metformin | Total
Number analyzed (Participants) | 177 | 162 | 169 | 508
Age, Continuous [Mean (Full Range); unit: years] | 57.3 [26 to 75] | 57.6 [18 to 75] | 56.8 [37 to 77] | 57.2 [18 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 88 | 101 | 282
  Male | 84 | 74 | 68 | 226
Body Weight [Mean (Standard Deviation); unit: kilograms] | 86.1 (15.6) | 84.2 (16.2) | 83.9 (13.9) | 84.8 (15.27)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: milligrams per deciliter] — Fasting Plasma Glucose
  milligrams per deciliter | 193.5 (52.4) | 194.6 (48.5) | 188.6 (49.7) | 192.2 (50.23)
HbA1c [Mean (Standard Deviation); unit: percentage] — Glycated hemoglobin measurement
  percentage | 8.9 (0.95) | 8.9 (0.94) | 9.0 (0.97) | 8.9 (0.95)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Change From Baseline for HbA1c Between TI+ Metformin and Metformin+Secretagogue
Time Frame: Baseline to Week 12
Population: Intention to Treat (ITT) Population with Last Observation Carried Forward
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of total hemoglobin
Groups:
- Metformin & Secretagogues: Metformin & Secretagogues
- TI Inhalation Powder + Metformin: Technosphere® Insulin Inhalation Powder & Metformin
Arm/Group | Metformin & Secretagogues | TI Inhalation Powder + Metformin
Number analyzed (Participants) | 162 | 169
Percentage of total hemoglobin | -0.78 (-0.78) [-0.92 to -0.64] | -0.70 (-0.70) [-0.84 to -0.56]
Statistical Analysis 1: Comparison: Metformin & Secretagogues vs TI Inhalation Powder + Metformin; ANCOVA fitting model change from baseline in A1c with fixed effects for treatment and pooled site and baseline A1c as a covariate; Test type: Superiority or Other; p = 0.420, ANCOVA; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.11 to 0.27]

2. Secondary Outcome: Difference in Change From Baseline for HbA1c Between TI Alone and Metformin+Secretagogue
Description: (Change from baseline within TI Alone) minus (change from baseline within metformin + secretagogue)
Time Frame: Baseline to Week 12
Population: Intention to Treat (ITT) Population for patients with available data
Measure: Mean (Standard Deviation); unit: Percentage of total hemoglobin
Groups:
- TI Inhalation Powder Alone: Technosphere® Insulin Inhalation Powder
Arm/Group | TI Inhalation Powder Alone | Metformin & Secretagogues
Number analyzed (Participants) | 133 | 153
Percentage of total hemoglobin | 0.12 (1.3) | -0.76 (0.92)
Statistical Analysis 1: Comparison: TI Inhalation Powder Alone vs Metformin & Secretagogues; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Type III; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [0.69 to 1.14]

3. Secondary Outcome: Change in HbA1c From Baseline to Week 24 (Subjects Who Stayed on Original Treatment)
Time Frame: Week 24
Population: Intent to Treat: Subjects who stayed on original treatment
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Arm/Group | TI Inhalation Powder Alone | Metformin & Secretagogues | TI Inhalation Powder + Metformin
Number analyzed (Participants) | 29 | 72 | 77
percentage of total hemoglobin | -1.82 (1.114) | -1.23 (1.080) | -1.68 (1.014)

ADVERSE EVENTS:
Time Frame: From first dose until 30 days after last dose of study medication
Description: Subjects in the TI Alone and Metformin + Secretagogue arms may have transferred to the TI + Metformin Arm for study period 2. There are 181, 166 and 351 subjects in the TI Alone, Metformin + Secretagogue and TI + Metformin treatment arms, respectively, across all 24 weeks of the study.
Arm/Group | TI Inhalation Powder Alone | Metformin & Secretagogues | TI Inhalation Powder + Metformin
Serious Adverse Events (participants affected / at risk) | 5/181 | 5/166 | 11/351
Other Adverse Events (participants affected / at risk) | 72/181 | 42/166 | 138/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TI Inhalation Powder Alone (N=181) | Metformin & Secretagogues (N=166) | TI Inhalation Powder + Metformin (N=351)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 0 | 1
ANGINA UNSTABLE (Cardiac disorders) | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 2 | 0
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 0 | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 1
CHOLECYCTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 1
SEPSIS (Infections and infestations) | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 2
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0 | 0
IIIRD NERVE PARALYSIS (Nervous system disorders) | 0 | 0 | 1
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 0 | 1 | 0
CALCULUS BLADDER (Renal and urinary disorders) | 0 | 0 | 1
URETHRAL STRICTURE (Renal and urinary disorders) | 0 | 1 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TI Inhalation Powder Alone (N=181) | Metformin & Secretagogues (N=166) | TI Inhalation Powder + Metformin (N=351)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 12 | 8
NASOPHARYNGITIS (Infections and infestations) | 4 | 13 | 18
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 24 | 21 | 84
COUGH (Respiratory, thoracic and mediastinal disorders) | 49 | 6 | 62

LIMITATIONS AND CAVEATS:
Wks 12-24 was a non-randomized treatment period of the trial; outcomes were not analyzed for Wks 12-24. Safety results include entire trial; patients counted in multiple treatments for safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the Study results subject to MNKD rights herein.